CLINICAL TRIAL: NCT00848913
Title: Effect of Rehabilitation With Versus Without Progressive Strength Training Implemented in the Acute Ward After Hip Fracture Surgery: A Randomized Controlled Trial
Brief Title: Strength Training After Hip Fracture Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hvidovre University Hospital (Other)
Responsible Party: Principal Investigator, Morten Tange Kristensen, Seniorresearcher, PhD, Hvidovre University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H-A-2007-0127 + 37036
Record Dates: First submitted 2009-02-19; First posted 2009-02-20 (Estimated); Last update posted 2015-06-03 (Estimated); Status verified 2015-06

CONDITIONS: Hip Fracture
Keywords: strength deficit; physical function
MeSH Terms: conditions — Hip Fractures | interventions — Rehabilitation; Resistance Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Rehabilitation without strength training (Active Comparator): Basic mobility and exercise therapy without strength training following a guideline with 12 specific exercises, progressed individually.
  Interventions: Other: Rehabilitation without strength training
- Rehabilitation with strength training (Experimental): Basic mobility and exercise therapy following a guideline with 12 specific exercises, progressed individually, and supplemented with progressive knee-extension strength training (10RM) of fractured limb every day during admission.
  Interventions: Other: Rehabilitation with strength training

INTERVENTIONS:
Other: Rehabilitation with strength training — Basic mobility and exercise therapy following a guideline with 12 specific exercises, progressed individually, and supplemented with progressive knee-extension strength training (10RM) of the fractured limb using ankle weight cuffs, daily during hospital stay.
  Arms: Rehabilitation with strength training
Other: Rehabilitation without strength training — Basic mobility and exercise therapy without strength training following a guideline with 12 specific exercises, progressed individually.
  Arms: Rehabilitation without strength training

SUMMARY:
The purpose of this study is to examine the effect of progressive strength training of the fractured limb in patients with hip fracture, during admittance in an acute orthopedic ward. The primary study hypothesis is that the training will reduce the strength deficit in the fractured limb in comparison with the non-fractured limb. Secondary, that patients following the intervention will present larger improvements in physical function compared to controls.

ELIGIBILITY:
Inclusion Criteria:

* Primary hip fracture surgery
* 65 years or older
* Speak and understand the Danish language
* Able to give informed consent
* Home-dwelling with and independent prefracture indoor walking ability equal to New Mobility Score >=2

Exclusion Criteria:

* Multiple fractures
* Weightbearing restrictions
* Patient unwilling to participate in appropriate rehabilitation
* Not able to cooperate to tests
* Terminal illness
* Patients who want an observer present at the information interview, but where such one is not available.
* Patients with a cervical hip fracture treated with Total Hip Arthroplasty or hip pins, due to expected short length of hospital stay.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 90 (Actual)
Dates: Start 2013-10; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Knee-extension strength in the fractured limb in comparison with the non-fractured limb. | At inclusion, at postoperative day 10 and/or at discharge.
  Maximal isometric knee-extension strength in the fractured limb in percentage of non-fractured limb. Isometric knee-extension strength will be measured using an externally fixated handheld dynamometer (Power Track II Commander; JTech Medical, Utah). A stap will be attached to the bed/chair and the patient's ankle (perpendicular to the lower leg), ensuring 90 degrees of knee flexion and an isometric contraction. The transducer will be placed under the strap at ankle level, just proximal to the malleolus, and the participant will be asked to extend the leg as forcefully as possible. Knee-extension strength will be expressed as the maximal voluntary torque per kilo body mass ([NIm]/kg), using the distance between the lateral femoral epicondyle and the center of the transducer and the body mass of each patient. The best of 4 trials for each limb will be used in analyses. The primary analysis will follow the intention-to-treat principle (last observation carried forward).

SECONDARY OUTCOMES:
Timed up and go test | From inclusion to postoperative day 10 and/or discharge
  Timed Up and Go test is assessed as early as possible during in-hospital stay and at discharge.

OTHER OUTCOMES:
10 meter fast speed, Cumulated Ambulation Score. | At discharge and during in-hospital stay.
  Cumulated Ambulation Score is recorded every day from inclusion to discharge. 10 meter fast speed is assessed at postoperative day 10 and/or discharge.
Short Falls Efficacy Scale-International (Short FES-I) | At discharge
  A questionnaire evaluation of the patient's subjective concern at the moment for falling related to 7 different physical functions. Score 7-28, with maximum score expressing very high concern of falling in all 7 physical functions.
Verbal Ranking Scale (VRS) | During in-hospital stay.
  Evaluation of experienced hip-fracture related pain at rest and during strength training and testing.
24-hour activity | From inclusion to discharge
  24-hour sit/lie and stand/walk activity measured by a ActivPAL3 activity monitor (PAL Technologies Ltd, Scotland) attached to the patient's non-fractured thigh.

CONTACTS AND LOCATIONS:
Overall Officials: Lise Kronborg, MSc, Principal Investigator — PMR-C, Copenhagen University at Hvidovre Hospital.
Locations (1):
- Department of Orthopedic Surgery hvidovre hospital, Hvidovre, Copenhagen, Denmark

REFERENCES:
- [Derived] Kronborg L, Bandholm T, Palm H, Kehlet H, Kristensen MT. Effectiveness of acute in-hospital physiotherapy with knee-extension strength training in reducing strength deficits in patients with a hip fracture: A randomised controlled trial. PLoS One. 2017 Jun 29;12(6):e0179867. doi: 10.1371/journal.pone.0179867. eCollection 2017. PMID 28662153